CLINICAL TRIAL: NCT02048423
Title: An Open Prospective Trial of IV Ketamine in Suicidal Adolescents
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00445
Record Dates: First submitted 2013-08-02; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Major Depressive Disorder
Keywords: suicidal
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental): Drug
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — IV Ketamine, 0.5 mg/kg X 15 mins. in PACU
  Other Names: Ketaset; Ketalean; Rogarsetic

SUMMARY:
1. Investigate the safety and effectiveness of a single dose of IV Ketamine for adolescents with suicidal ideation and depression. It is hypothesize that Ketamine will be well tolerated and significantly reduce depressive symptoms and suicidal ideation.
2. Explore whether decision making as measured by the Iowa Gambling Task changes before and after Ketamine infusion. It is hypothesize that IV Ketamine infusion will significantly improve the decision making ability a measured by the Iowa Gambling Task in adolescents that are suicidal.

DETAILED DESCRIPTION:
This is an open prospective study of a single, low dose (0.5 mg/kg) intravenous (IV) Ketamine in 10 adolescent subjects admitted to Nationwide Childrens Hospital following a serious suicide attempt and who meet criteria for major depression or bipolar disorder I, current episode depressed. Subjects will be recruited via the psychiatry consult service, evaluated on the floor and if eligible and consent is obtained, transferred to the PACU for IV Ketamine infusion. Following infusion and when PACU discharge criteria are met, subjects will be transferred back to their floor for medical and psychiatric monitoring until they can be transferred to an inpatient psychiatric unit for additional care. Subjects will be transferred to an inpatient psychiatric unit for continued psychiatric care as part of their routine psychiatric care via the consult team. The research team will follow-up by telephone one week and four weeks after Ketamine injection to collect additional information about the patient's overall course and response.

ELIGIBILITY:
Inclusion Criteria

* Subjects age 12 years 0 months to 17 years, 11 months old
* Voluntary admission for a suicide attempt requiring medical intervention in the previous 24-48 hours (Kiddie Schedule for Affective Disorders Suicide Behavior Score > 3).
* Meets criteria for major depression, single- or recurrent episode, non-psychotic or Bipolar I, current episode depressed, with a baseline Inventory for depression score of > 16.
* The patient and legal guardian must understand the nature of the study and be able to comply with protocol requirements. The legal guardian must give written informed consent and the youth, written assent.
* English is spoken as the primary language in the home.

Exclusion Criteria

* Any serious, unstable medical illness or clinically significant abnormal laboratory assessments that would adversely impact the scientific interpretability or unduly increase the risks of the protocol.
* Admitted to Nationwide Children's Hospital involuntarily.
* Unable to assent because of severe mental retardation or incapacitating psychosis.
* Other medications: See Table 1. The list in Table 1 is not exhaustive. The Principal Investigator and the Co-Investigator will review all concomitant medicines and any medicine that could interfere with the trial will be considered exclusionary. Subjects with bipolar disorder will be allowed to continue their mood stabilizers and or antipsychotic agents at the discretion of the investigator. Stimulants use is acceptable, though the child must be on a stable dose for the past 3 months and the dose must not be changed through the trial. A stable dose is defined as no more that 25% change in the total daily dose of a stimulant.
* General medical conditions: children with major medical conditions that would interfere with involvement in the study or the study medication will not be enrolled.
* Exclusionary Psychiatric Conditions: Autism, substance dependence, psychosis or psychotic major depression.
* History of physical, sexual, or emotional abuse, which results in a clinically significant impact on clinical presentation, potentially driving some of the symptoms of major depressive disorder.
* Receipt of an investigational drug within 30 days prior to study entry.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in Quick Inventory of Depression Clinician (QIDS-C) total scores from baseline to endpoint and Clinical Global Improvement Score. | 2 days

SECONDARY OUTCOMES:
Clinical Global Assessment Scale | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Kowatch, MD, PhD, Principal Investigator — OSU Medical Center/Nationwide Childrens Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States